CLINICAL TRIAL: NCT01993407
Title: Training Executive Functions to Facilitate Recovery Following Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: New Jersey Commission on Brain Injury Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-743-12
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Traumatic Brain Injury; Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Task Switching Training (Experimental): Participants will complete four, one-hour training sessions in which they will practice switching between tasks within an alternating runs task switching paradigm.
  Interventions: Behavioral: Task Switching Training
- Pure Task Training (Placebo Comparator): Participants will complete four, one-hour training sessions in which they will perform a single task each session, alternating tasks between but not within sessions.
  Interventions: Behavioral: Control Task

INTERVENTIONS:
Behavioral: Task Switching Training — Participants will complete four, one-hour training sessions in which they will practice switching between tasks within an alternating runs task switching paradigm.
  Arms: Task Switching Training
Behavioral: Control Task — Participants will complete four, one-hour training sessions in which they will perform a single task each session
  Arms: Pure Task Training

SUMMARY:
The purpose of this research study is to investigate different types of task training to determine if training improves thinking processes following traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* If you have had a Traumatic Brain Injury (TBI)or no history of neurological disease/damage.
* If you are between the ages of 19 and 65.

Exclusion Criteria:

For participants with Traumatic Brain Injury:

* If you have a history of prior neurological disorders (e.g., stroke, seizures, or brain tumor).
* If your Brain injury is less than 6 months ago.

For healthy participants:

-If you have a history of prior neurological disorders (e.g., head injury, stroke, seizures, or brain tumor).

For All participants:

* If you have significant psychiatric history (such as schizophrenia or bipolar disorder.)
* If you have a alcohol or drug abuse history.
* If you are currently taking certain types of medications, which the study doctor will review.
* If you do not have a working knowledge of the English Language.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in switch costs, measured via response time in milliseconds on task switch trials minus response time on task repetition trials, from baseline | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Starla Weaver, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation Research Center, West Orange, New Jersey, United States